CLINICAL TRIAL: NCT03737084
Title: Effects of the Cognitively-Based Compassion Training (CBCT) Adapted to Patients Undergoing Hematopoietic Stem Cell Transplant (HSCT) and Their Caregivers on Biological and Psychosocial Parameters
Brief Title: Effects of Compassion Training to Patients Undergoing HSCT on Biological and Psychosocial Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEP 2.373.269
Record Dates: First submitted 2018-10-29; First posted 2018-11-09 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: hematopoietic stem cell transplant; cancer; compassion; meditation; depression; anxiety; heart rate variability; resilience
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group: The compassion intervention (CBCT) will be performed during the period of hospitalization, in the hospital room, and will be applied simultaneously to the patient his caregiver.
  Control Group: Patients and caregivers in the control group will receive standard hospital care. Patients and caregivers of the control group will receive the same compassion intervention at the end of the study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBCT Intervention (Experimental): The compassion intervention (CBCT) will be performed during the period of hospitalization, in the hospital room, and will be applied simultaneously to the patient his caregiver. The training consists of six weekly sessions. The participant will receive six guided meditation audio, relative to each session, to practice during the week.
  Interventions: Behavioral: CBCT Intervention
- Control group (No Intervention): Control group participants will receive standard hospital care. Patients and caregivers of the control group will receive the same CBCT intervention at the end of the study.

INTERVENTIONS:
Behavioral: CBCT Intervention — The training consists of six weekly sessions. The participant will receive six guided meditation audio, relative to each session, to practice during the week.
  Arms: CBCT Intervention

SUMMARY:
The hematopoietic stem cell transplant (HSCT) experience is emotionally and physically stressful for cancer patients who undergo this procedure. This study aims to evaluate the effects of Cognitively-Based Compassion Training (CBCT) on depression and anxiety symptoms, levels of resilience, hope and self-compassion in patients undergoing HSCT and their caregivers. As well as assessing the effects of CBCT on clinical conditions in patients and cortical activity and heart rate variability in caregivers.

DETAILED DESCRIPTION:
The study hopes to show the positive effects of compassion training in patients and their caregivers.

Overall aim:

This study aims to evaluate the effects of Cognitively-Based Compassion Training (CBCT) on: depression and anxiety symptoms; levels of hope; resilience; mindfulness; self-compassion and quality of life. The study also aims to demonstrate whether CBCT training has any effect on clinical parameters of transplanted patients, as well as whether it has an effect on cortical activity and heart rate variability inpatients and caregivers.

Specific objectives:

1. Develop an adaptation of the CBCT protocol for hospitalized patients;
2. To evaluate the effect of CBCT on depressive and anxious symptoms in patients and their caregivers;
3. To evaluate the effect of CBCT on resilience, quality of life and self-compassion in patients and their caregivers;
4. Investigating the CBCT training results in altering the cortical activity of patients and caregivers while performing a recall task of recent autobiographical experiences;
5. Investigate whether CBCT training results in changes in heart rate variability in patients and caregivers;
6. To investigate whether CBCT training has any effect on patient's levels of symptoms, such as: pain, nausea, insomnia, among others;
7. To evaluate how correlations between psychosocial factors and biological markers: cortical activity and heart rate variability;
8. Evaluate perceptions and impressions of patients and caregivers on the protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for HSCT attended at Albert Einstein Hospital, as well as their respective caregivers.

Exclusion Criteria:

* history of severe psychiatric disorders and neurological diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Anxiety and Depression symptoms at 1 week after intervention | baseline,1 week after intervention
  Hospital Anxiety and Depression Scale (HADS). The scale consists of 14 items, 7 for anxiety (HADS-A) and 7 items for depression (HADS-D). The final score ranges from 0 to 21 points in each subscale, the higher the score, the greater the symptoms of anxiety or depression (Zigmond and Snaith, 1983).
Change from Baseline Resilience level at 1 week after intervention | baseline; 1 week after intervention.
  Resilience Scale (RS). Developed by Wagnild and Young (Wagnild and Young, 1993). Composed of 25 items. The Resilience Scale was applied to measure the degree of resilience. It measures two main factors: 'personal competence' (17 items) and 'acceptance of self and life' (8 items). The response scale ranges from 1 ('totally disagree') to 7 ('totally agree'). The total score ranges from 26 to 175 points. The higher the score the higher the level of resilience.
Change from Baseline Self-Compassion level at 1 week after intervention | baseline; 1 week after intervention.
  Self-Compassion Scale. This is a 26-item scale that measures how one typically acts toward oneself in difficult times. These items were designed to assess how respondents perceive their actions toward themselves in difficult times and are rated using a Likert-type scale anchored from 1 (almost never) to 5 (almost always). The scale ranges from 26 to 130 points. The higher the score the higher the level of Self-Compassion. Developed by Kristin Neff.
Change from Baseline Perceived Stress level at 1 week after intervention | baseline; 1 week after intervention.
  Perceived Stress Scale (PSS). This scale measures the degree to which individuals perceive situations as stressful. Composed of 14 items related to sensation. PSS scores are obtained by reversing the scores on the seven positive items, e.g., 0=4, 1=3, 2=2, etc., and then summing across all 14 items. Items 4, 5, 6, 7, 9, 10, and 13 are the positively stated items. A higher score indicates a higher level of Perceived Stress. The final score ranges from 0 to 56 points. Developed by Luft, 2007.

OTHER OUTCOMES:
Cortical activity | baseline, 1 week after intervention
  Measured by Near-Infrared Spectroscopy (NIRS), in an experiment using a paradigm of autobiographical events, remembering stressful and positive memories.
Heart rate variability (HRV) | baseline, 1 week after intervention
  Measured from the cardiac activity record through a Polar® V800 heart monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Kozasa, PhD, Principal Investigator — Instituto Israelita de Ensino e Pesquisa Albert Einstein
Locations (2):
- Brazil (2):
  - Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo

REFERENCES:
- [Background] Kozasa EH, Radvany J, Barreiros MA, Leite JR, Amaro E Jr. Preliminary functional magnetic resonance imaging Stroop task results before and after a Zen meditation retreat. Psychiatry Clin Neurosci. 2008 Jun;62(3):366. doi: 10.1111/j.1440-1819.2008.01809.x. No abstract available. PMID 18588603
- [Background] Dodds SE, Pace TW, Bell ML, Fiero M, Negi LT, Raison CL, Weihs KL. Feasibility of Cognitively-Based Compassion Training (CBCT) for breast cancer survivors: a randomized, wait list controlled pilot study. Support Care Cancer. 2015 Dec;23(12):3599-608. doi: 10.1007/s00520-015-2888-1. Epub 2015 Aug 16. PMID 26275769